CLINICAL TRIAL: NCT05606887
Title: Investigating Proactive, Digital Methods to Identify Signs and Symptoms of Mental Health Distress in Emergency Medicine Physicians
Brief Title: Identifying Mental Health Distress in EM Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0852220
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional | interventions — Wearable Electronic Devices; Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the intervention arm (with wearable devices or EMAs) or control (survey-only) in parallel and will remain in their assigned arm throughout their participation in the survey.
Masking Description: Given the nature of the intervention (i.e., participants in the intervention arm receiving a wearable device and investigators and analysts reviewing biometric data for this group), the study will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to completing 3 surveys over the course of 6 months, participants in the intervention arm will be asked to wear a wearable device (FitBit Charge 5), complete texting-based ecological momentary assessments to gauge real-time feelings of stress, and receive bi-weekly personalized data dashboards to report back their data.
  Interventions: Other: Wearable Device and Ecological Momentary Assessments
- Control (No Intervention): Participants randomized to this arm will receive digital surveys over the course of 6 months (one at baseline, one at 3 months, and one at 6 months). These surveys will be the same as the intervention arm and will ask questions related to burnout, anxiety, depression, PTSD, and stress.

INTERVENTIONS:
Other: Wearable Device and Ecological Momentary Assessments — The intervention will consist of three components:
  1. Completion of brief text-message based surveys 2-3 times per week
  2. Wearing a wrist-based wearable device to generate individual data insights on physiological data related to stress and well-being, including heart rate variability, stress scores, and sleep quality
  3. Individual biweekly reports of survey response trends and curated resources intended to support participant well-being
  Arms: Intervention

SUMMARY:
This project seeks to develop and test provider-centered strategies that improve the detection and facilitate the treatment of physiologic and mental health symptoms in emergency medicine physicians. This will be done by investigating the feasibility and acceptability of wearable device and EMA feedback with personalized linkage to an evidence-based mental health platform at the University of Pennsylvania Health System.

DETAILED DESCRIPTION:
This proposal aims to conduct a 3-month pilot randomized control trial (n=60) testing feasibility, acceptability, and the exploratory effectiveness of digital data feedback (wearables and EMA) with tailored, symptom-specific linkage to mental health and resilience resources versus control on mental health symptoms (depression, anxiety, PTSD) and burnout in EM clinicians. The study will recruit and enroll 60 emergency medicine physicians, residents, and advanced practice providers via email and inperson outreach. Once enrolled, both arms be asked to take a baseline survey which will measure their level of well-being, burnout, depression, and anxiety.

Study participants will be randomized following consent and completion of baseline surveys. Participants will be randomly assigned to usual care or intervention. We will use 2:1 randomization. We will randomize in block sizes of 3 and 6.

Intervention: The intervention arm will then be given a wearable device and will be asked to wear it for 3 months. The device will collect biometric data on stress levels, sleep patterns, and other physiological measures of well-being. The intervention group will receive biweekly EMA short surveys, personalized bi-weekly reports from their EMA data, biometric feedback from wearable devices (sleep, heart rate variability, physical activity), and linkage to tailored and symptom-specific Cobalt resources on health and resilience. After 3 months, we will survey providers to complete a post-survey followed by a survey at 6-months following a 3-month washout period.

Control: The control arm will be asked to complete a baseline survey as well as one assessment at the end of the three-month study period. They will receive usual care, or clinician-initiated use of Penn Cobalt. They will then complete additional surveys at 3-months and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Emergency Medicine (EM) physician or advanced practice provider
* Daily access to smart phone
* Ability to use a wrist-worn wearable device
* Has or is willing to create a Gmail / Google account
* Provides at least 20 hours per week of clinical care.

Exclusion Criteria:

* Under 18
* Not a Penn EM physician or advanced practice provider
* Does not have daily access to a smart phone
* Unwilling or unable to wear a wearable device
* Does not have or is unwilling to create a Gmail / Google account
* Does not provide at least 20 hours per week of clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention (FIM) | Through study completion, on average 6 months
  Feasibility will be measured by the Feasibility of Intervention Measure (FIM)
Feasibility of Intervention (Study Retention) | Through study completion, on average 6 months
  Feasibility will be measured by study retention
Acceptability of Intervention (AIM) | Through study completion, on average 6 months
  Acceptability will be measured by the validated Acceptability of Intervention Measure.
Acceptability of Intervention (EMA Completion Rates) | Through study completion, on average 6 months
  Acceptability will be measured by the open/completion rates of ecological momentary assessment.

SECONDARY OUTCOMES:
Anxiety | Through study completion, on average 6 months
  While the study will not be powered to detect effectiveness of the device on stress and other mental health indicators, secondary outcome measures will explore the potential for effect. The GAD-7 will be used to measure anxiety.
Depression | Through study completion, on average 6 months
  While the study will not be powered to detect effectiveness of the device on stress and other mental health indicators, secondary outcome measures will explore the potential for effect. The PHQ-8 will be used to measure depression.
Professional Burnout | Through study completion, on average 6 months
  While the study will not be powered to detect effectiveness of the device on stress and other mental health indicators, secondary outcome measures will explore the potential for effect. The Stanford Professional Fulfillment Index will be used to measure burnout.
Post-Traumatic Stress Disorder | Through study completion, on average 6 months
  While the study will not be powered to detect effectiveness of the device on stress and other mental health indicators, secondary outcome measures will explore the potential for effect. The PC-PTSD-5 will be used to measure PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No